CLINICAL TRIAL: NCT05901051
Title: Randomized and Controlled Clinical Study of High-dose Dual Therapy with Different Administration Frequencies in the Treatment of Helicobacter Pylori
Brief Title: High-dose Dual Therapy with Different Administration Frequencies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjyy20210815
Record Dates: First submitted 2023-02-24; First posted 2023-06-13 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Dual Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dual therapy A (Experimental): Vonoprazan 20mg bid ac and amoxicillin 0.75g qid pc
  Interventions: Drug: vonoprazan; Drug: Amoxicillin
- dual therapy B (Experimental): Vonoprazan 20mg bid ac and amoxicillin 1g tid pc
  Interventions: Drug: vonoprazan; Drug: Amoxicillin
- dual therapy C (Experimental): Vonoprazan 20mg bid ac and amoxicillin 1g tid ac
  Interventions: Drug: vonoprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: vonoprazan — Potassium competitive acid blocker
Drug: Amoxicillin — Antibiotics for H. pylori eradication

SUMMARY:
This study is a single center, randomized controlled clinical study. The enrolled patients are HP positive. They are diagnosed as HP positive by rapid urease test and/or 13C urea breath test. According to the declaration of Helsinki, 327 patients will be included in this study. After obtaining the written informed consent of the patients, HP culture and drug sensitivity test will be conducted on all the selected patients with the success rate, adverse reactions, compliance, antibiotic resistance of HP and its impact on HP eradication.

DETAILED DESCRIPTION:
According to relevant literature research, amoxicillin TID groups (including before meal group and after meal group) were given Vonorasen (Takeda China) 20mg bid and Amoxicillin 1.0 TID (Zhejiang Jinhua Kangenbei biopharmaceutical Co., Ltd.). Amoxicillin Qid group was given Vonorasen (Takeda China) 20mg bid and Amoxicillin 0.75 Qid (Zhejiang Jinhua Kangenbei biopharmaceutical Co., Ltd.), all the drugs were purchased by the patients from the hospital. The three groups were treated for 14 days respectively, and 13C urea breath test was performed 6 weeks after drug withdrawal. The negative ones were judged as HP eradication.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection

Exclusion Criteria:

* Pregnant and lactating women;
* History of gastrointestinal malignancies;
* History of previous subtotal gastrectomy;
* Serious dysfunction of heart, liver, kidney, lung and other important organs and congenital diseases; Such as grade IV cardiac insufficiency, liver failure, uremia, respiratory failure, hemophilia, Wilson disease, etc;
* History of hematological diseases
* People who are allergic to drugs;
* The guardian or patient refused to join the group;
* Alcohol and / or drug abuse (addiction or dependence) or poor compliance judged by doctors;
* No legal capacity or poor self-knowledge
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 8 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-rea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse events | Within 7 days after completion of therapy
  The subjects were asked to record side effects and discomfort during treatment and actual drug administration.
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu S, Huang Y, Chen J, Guo Y, Li M, Ding Z, Liang X, Lu H. Vonoprazan-Amoxicillin Dual Therapy With Different Amoxicillin Administration Regimens for Helicobacter pylori Treatment: A Randomized Controlled Trial. Helicobacter. 2024 Jul-Aug;29(4):e13118. doi: 10.1111/hel.13118. PMID 39087868